CLINICAL TRIAL: NCT07124234
Title: Assessment of the Impact of Social Anxiety on Primary Headache in Adolescents: A Case-Control Study
Brief Title: The Impact of Social Anxiety on Adolescents Diagnosed With Primary Headache: A Case-control Study
Status: Not yet recruiting | Type: Observational
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Fatma SARGIN, M.D, MD, Konya Necmettin Erbakan Üniversitesi
Other Study IDs: 2025001
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Primary Headache; Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Participants who will be diagnosed with primary headache according to InternationalClassification of Headache Disorders, 3rd edition (ICHD-3) criteria, confirmed by a pediatric neurologist
- Control group: Participants who will have no history of recurrent headache or chronic physical/psychiatricillness

SUMMARY:
This case-control study will examine whether adolescents aged 12-18 years with a diagnosis of primary headache are more likely to experience elevated social anxiety compared to matched healthy controls. Social anxiety will be assessed using the SAS-A, and the study will also explore whether environmental and sociodemographic factors such as tobacco smoke exposure, BMI, and parental education influence this relationship.

DETAILED DESCRIPTION:
The study will include adolescents aged 12-18 years who have been diagnosed with primary headachebased on the International Classification of Headache Disorders, 3rd edition (ICHD-3). The main exposure ofinterest will be the presence and severity of social anxiety, which will be measured using the Social AnxietyScale for Adolescents (SAS-A), a validated self-report questionnaire. The SAS-A takes approximately 10minutes to complete. Additional variables that will be collected will include sociodemographiccharacteristics, BMI, parental education levels, income status, parental smoking habits, and theadolescent's exposure to secondhand and thirdhand tobacco smoke. All assessments, includingquestionnaires and physical measurements (height and weight), are expected to be completed inapproximately 20 minutes per participant. The total observation duration for each participant will be about30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18 years
* Case group: Participants who will be diagnosed with primary headache according to InternationalClassification of Headache Disorders, 3rd edition (ICHD-3) criteria, confirmed by a pediatric neurologist
* Control group: Participants who will have no history of recurrent headache or chronic physical/psychiatricillness

Exclusion Criteria:

* History of neurological disease other than primary headache
* Any previously diagnosed psychiatric disorders
* Regular use of psychotropic medications
* Cognitive or developmental disabilities that would interfere with assessments

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Case group: Participants who will be diagnosed with primary headache according to InternationalClassification of Headache Disorders, 3rd edition (ICHD-3) criteria, confirmed by a pediatric neurologist Control group: Participants who will have no history of recurrent headache or chronic physical/psychiatricillness
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Total score on the Social Anxiety Scale for Adolescents (SAS-A) | Day 1
  The SAS-A, a self-administered 22-item Likert-scale questionnaire

SECONDARY OUTCOMES:
Prevalence of clinically significant social anxiety (SAS-A = 50) | Day 1
  Classification based on SAS-A total score cut-off
Body Mass Index (BMI) differences between groups | Day 1
  BMI calculated as kg/m²
Parental smoking status | Day 1
  Self-report from caregiver; statistical comparison of SAS-A scores by smoking exposure

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data
Supporting Information: CSR
Access Criteria: Requires review on a case-by-case basis by the trial custodian, sponsor or data sharing committee
  • Requires a scientifically sound proposal or protocol
  • Requires approval by an ethics committee
  • Requires a data sharing agreement between data requester and trial custodian or sponsor